CLINICAL TRIAL: NCT01586780
Title: Effects of Pre-meal Drinks With Protein and Amino Acids on Glycemic and Metabolic Responses at a Subsequent Composite Meal
Brief Title: Metabolic Effects of a Pre-meal Protein Drink With or Without Added Amino Acids at a Subsequent Composite Meal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Principal Investigator, Ulrika Gunnerud, Msc, Post Graduate student, Lund University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: Dnr 1.556/2008
Record Dates: First submitted 2012-04-23; First posted 2012-04-27 (Estimated); Last update posted 2012-04-27 (Estimated); Status verified 2012-04

CONDITIONS: Diabetes Mellitus, Type 2; Satiety Response
Keywords: Whey protein; Soy protein; Insulinogenic amino acids; Incretins; Glycaemia; Insulinaemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (7):
- Reference meal (Experimental)
  Interventions: Dietary Supplement: Reference meal
- Whey protein (Experimental)
  Interventions: Dietary Supplement: Protein drink
- Whey + 5 amino acids (Experimental)
  Interventions: Dietary Supplement: Protein drink
- Whey + 6 amino acids (Experimental)
  Interventions: Dietary Supplement: Protein drink
- Soy protein drink (Experimental)
  Interventions: Dietary Supplement: Protein drink
- Soy + 5 amino acids (Experimental)
  Interventions: Dietary Supplement: Protein drink
- Soy + 6 amino acids (Experimental)
  Interventions: Dietary Supplement: Protein drink

INTERVENTIONS:
Dietary Supplement: Protein drink — Test drink providing 9g protein
  Arms: Soy + 5 amino acids; Soy + 6 amino acids; Soy protein drink; Whey + 5 amino acids; Whey + 6 amino acids; Whey protein
Dietary Supplement: Reference meal — Control meal
  Arms: Reference meal

SUMMARY:
The purpose of the study was to investigate the efficacy of intake of whey or soy protein isolates, respectively, with or without supplementation of amino acids, on post-meal insulin secretion and glycaemic regulation. Additionally, the effect on plasma amino acids, gut hormones and ghrelin in plasma, as well as subjective satiety was investigated.

DETAILED DESCRIPTION:
Hyperglycaemia in type 2 diabetes (T2D) is associated with an increased risk of cardiovascular diseases, and it has been suggested that reduction of postprandial glycaemia is just as important as lowering fasting blood glucose levels to reach optimal metabolic control and reduce risk of complications in T2D. Observational studies indicate that milk consumption reduces the risk of developing T2D, obesity and cardiovascular disease, and a possible protective mechanism has been ascribed to the protein fraction. It has previously been demonstrated that addition of whey proteins, co-ingested with carbohydrates, stimulates insulin secretion and reduces postprandial glycaemia in both healthy subjects as well as in T2D patients. The effect is mediated through the insulinogenic properties of whey that appears to stem from a generation of a particular amino acid (AA) pattern in postprandial blood after ingestion of whey proteins. In the presently described project it is hypothesized that exchanging part of the whey protein for insulinogenic AA might be useful to optimize an insulinogenic effect. Additionally, soy protein has been suggested to have beneficial effects on insulin resistance and obesity as well on satiety. The possible effect of soy protein on insulin response and glycaemic regulation is therefore also of interest.

A randomized, single blind, within-subject trial was performed. The test meals were provided as breakfasts on 7 different occasions in random order with approximately 1 week between each test. The test subjects were instructed to drink the protein drink immediately prior to eating the standardized sandwich meal. Altogether, the protein drink and the sandwich meal were to be consumed within 12 min.

ELIGIBILITY:
Inclusion Criteria:

* normal fasting blood glucose
* normal BMI

Exclusion Criteria:

* smokers
* vegetarians
* subjects who receives any drug treatment
* lactose malabsorption

Ages: 20 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2009-08; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Blood glucose, insulin, amino acids, ghrelin and incretins | Acute postprandial phase (0-180 min)

SECONDARY OUTCOMES:
Subjective satiety | 3h postprandial (0-180 min)

CONTACTS AND LOCATIONS:
Overall Officials: Inger Björck, Professor, Study Chair — Lund University; Ulrika Gunnerud, MSc, Principal Investigator — Lund University
Locations (1):
- Applied Nutrition and Food Chemistry, Lund University, Lund, Sweden

REFERENCES:
- [Derived] Gunnerud UJ, Heinzle C, Holst JJ, Ostman EM, Bjorck IM. Effects of pre-meal drinks with protein and amino acids on glycemic and metabolic responses at a subsequent composite meal. PLoS One. 2012;7(9):e44731. doi: 10.1371/journal.pone.0044731. Epub 2012 Sep 19. PMID 23028596